CLINICAL TRIAL: NCT06865118
Title: The Nor-SSCardioCare Pilot Trial: Home-Based Clinical Management of Cardiac Complications in Systemic Sclerosis Patients
Brief Title: Home-Based Clinical Management of Cardiac Complications in Systemic Sclerosis
Acronym: Nor-SScCare
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anna-Maria Hoffmann-Vold, Prof Dr med, Oslo University Hospital
Other Study IDs: 762859
Record Dates: First submitted 2025-02-17; First posted 2025-03-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis (SSc); Pulmonary Arterial Hypertension (PAH); Home Monitoring Follow-up
Keywords: Systemic Sclerosis; Pulmonary arterial hypertension; Home monitoring; Remote monitoring; Observational study; PAH progression; Disease progression; Home-based markers
MeSH Terms: conditions — Scleroderma, Systemic; Pulmonary Arterial Hypertension; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SSc-PAH: This study includes adult patients diagnosed with systemic sclerosis-associated pulmonary arterial hypertension (SSc-PAH) who meet predefined eligibility criteria. All participants will undergo home monitoring using digital tools and attend two hospital visits for clinical assessments. The study aims to assess the feasibility, validity, and reliability of home-based monitoring in SSc-PAH patients. Participants will perform biweekly symptom reporting, functional tests, and blood sampling at home, in addition to comprehensive clinical evaluations at baseline and week 12. Home-based assessments will be compared to hospital-based assessments within the same participants to explore their agreement and potential clinical utility. The findings will inform the design of a future study on integrating home monitoring into routine clinical care.

SUMMARY:
The goal of this observational pilot trial is to evaluate the feasibility of home monitoring for patients with systemic sclerosis-associated pulmonary arterial hypertension (SSc-PAH). The study will assess home-based measures that may help detect disease progression earlier and will also evaluate patient satisfaction, usability, and the impact on health-related quality of life.

The study aims to answer:

* How feasible is home monitoring in SSc-PAH patients in terms of adherence, technical feasibility, and validity of home-based measures?
* How do home-based assessments compare to hospital-based assessments in detecting disease progression?
* How do patients experience digital home monitoring?

Participants will:

* Use a digital platform (Zeen Health) for biweekly self-reporting of symptoms and physiological measurements.
* Perform functional tests at home, including the 1-minute sit-to-stand test (1MSTS).
* Wear the ECG247 Smart Heart Sensor for one week to monitor heart rhythm.
* Collect and submit home blood samples every two weeks.
* Attend two hospital visits (baseline and week 12) for clinical assessments, functional testing, pulmonary function tests, echocardiography, and routine blood sampling for clinical assessments.

This 12-week study will assess the feasibility of home monitoring, as well as the validity and reliability of home-based measures. The findings will help design a future study aimed at integrating home-based assessments into routine clinical care.

DETAILED DESCRIPTION:
Study Overview The Nor-SSCardioCare Pilot Trial is a prospective, observational, single-arm feasibility study evaluating the implementation of home monitoring in patients with systemic sclerosis-associated pulmonary arterial hypertension (SSc-PAH).

The primary objective is to assess the feasibility of home monitoring in terms of patient adherence, technical feasibility, and the validity and reliability of home-based measures compared to hospital-based assessments.

Additionally, the study will evaluate patient satisfaction, usability of digital home monitoring, and its impact on health-related quality of life (HRQoL).

This 12-week study will generate feasibility data to inform the design of a larger trial aimed at integrating home monitoring into clinical care for earlier detection of disease progression and cardiac complications.

Background and Rationale SSc-PAH is a life-threatening complication of systemic sclerosis (SSc), with a high mortality rate and limited treatment response if diagnosed late.

Currently, disease progression may go undetected between hospital visits, as patients are typically seen every 3-6 months for assessments including: echocardiography, pulmonary function tests (PFTs), 6-minute walk distance (6MWD) test, right heart catheterization (RHC) when needed.

However, fixed-interval follow-ups do not always capture early signs of disease worsening. Digital home monitoring may improve disease management by allowing more frequent patient assessments (biweekly vs. standard hospital visits), earlier detection of PAH progression based on physiological and symptom data, and increased patient engagement and self-management.

The pilot trial will assess home-based measures that may contribute to earlier detection of disease progression, explore their validity and reliability compared to hospital-based assessments, and evaluate patient satisfaction, usability, and impact on health-related quality of life (HRQoL).

This 12-week study will generate feasibility data to inform the development of a larger trial focused on integrating home monitoring into clinical care.

Objectives and Endpoints

Primary Objective:

To evaluate the feasibility of home monitoring for SSc-PAH patients, including:

* Patient adherence and compliance (frequency and completeness of data entries, ECG monitoring compliance).
* Technical feasibility (rate of technical failures, data loss, and missing entries).
* Validity and reliability of home-based measures compared to hospital-based assessments (comparison of home-based 1MSTS vs. hospital-based 6MWD, and home-based NT-proBNP vs. hospital-based NT-proBNP).

Secondary Objectives:

* Evaluate patient satisfaction, usability, and HRQoL of home monitoring.
* Comparison of home-based vs. hospital-based risk stratification (e.g., mMRC vs. WHO functional class, home-based 1MSTS vs. hospital-based 1MSTS, and NT-proBNP).
* PAH progression and PAH events.
* Heart rhythm monitoring, including arrhythmia detection, heart rate variability (HRV), and its correlation with PAH severity.
* Reproducibility of home-based measures to assess reliability across different settings.

Exploratory analysis

• Explore biomarkers and their correlation with PAH severity

Study Design and Methods

Study Type:

* Prospective, observational, single-arm feasibility study.
* Study duration: 12 weeks.
* Sample size: 20 patients diagnosed with SSc-PAH.
* Study site: Conducted at Oslo University Hospital (OUH), Norway.

Study Procedures and Data Collection

This 12-week study will consist of:

* Two hospital visits at Oslo University Hospital (OUH) (baseline and week 12) for clinical assessments, including functional tests, pulmonary function tests (PFTs), echocardiography, routine blood sampling for clinical assessments, including NT-proBNP measurements, and reporting of patient-reported outcomes using validated HRQoL questionnaires (EmPHasis-10, ScleroID, EQ-5D-5L, HAQ, HADS) and patients satisfaction questionnaires (CSQ-8, Usability, Feasibility, and Impact Questionnaire).
* Biweekly home monitoring, where participants will report symptoms via a digital platform (Zeen Health), perform home-based functional tests (1-minute sit-to-stand test, 1MSTS), collect capillary blood samples for biomarker analyses and NT-proBNP, and undergo ECG monitoring for one week.

Quality Assurance and Data Validation

1. Data Entry and Validation

   * Zeen Health Platform: Secure, approved digital platform used for collecting real-time patient-reported data.
   * Regular monitoring of data completeness, technical issues, and adherence.
   * Manual cross-checks of selected entries against medical records for accuracy.
2. Registry Data Management

   * Secure data storage in Tjeneste for Sensitive Data (TSD) at the University of Oslo.
   * Data review meetings to ensure accuracy and completeness.
   * Consistency checks to verify alignment of registry data with predefined variables.
3. Data Dictionary and Coding Standards

   * Standardized variable definitions for home-based and hospital-based measures.
   * Data coded using predefined categories (e.g., WHO-FC classifications, NT-proBNP cutoffs).
4. Source Data Verification

   * Selected data will be cross-checked against hospital medical records.
   * Agreement between home-based and hospital-based assessments will be analyzed.
5. Sample Size Justification

   * 20-patient sample chosen to assess feasibility before scaling to a larger trial.
   * Not powered for clinical efficacy outcomes.
6. Plan for Missing Data

   * Patient reminders: Participants who miss scheduled data entries may receive gentle reminders via the digital platform to improve adherence.
   * Monitoring of missing data patterns: If systematic issues are identified, additional measures may be implemented.
   * No statistical imputation: Missing data will not be imputed but will be analyzed descriptively.

Statistical Analysis Plan

* Descriptive statistics (means, SDs, proportions) will be used for feasibility outcomes.
* Agreement analysis:

  * Bland-Altman plots for home-based 1MSTS vs. 6MWD.
  * Intraclass correlation coefficients (ICC) for home-based NT-proBNP vs. hospital-based NT-proBNP.
* HRQoL and usability outcomes will be analyzed using paired t-tests/Wilcoxon tests.
* Heart rhythm data (arrhythmia type/frequency, HRV) will be analyzed and correlated with PAH risk profiles.

Ethical Considerations and Oversight

* Approved by the Regional Committees for Medical and Health Research Ethics (REK Sør-Øst, Norway).
* Informed consent required before participation.
* No experimental therapies; all participants will receive standard clinical care.
* Patient confidentiality protected under GDPR compliance.

Future Directions Findings from this study will inform the design of a larger clinical trial evaluating whether home monitoring improves early detection of PAH progression and enhances patient outcomes. If successful, future research will assess its clinical utility in routine care and its potential for broader implementation in SSc-PAH management.

Potential benefits of a future trial:

* Cost-effective, remote disease monitoring.
* Earlier intervention for PAH worsening.
* Improved patient engagement and HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilment of the 2013 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) SSc classification criteria
* Fulfilment of the 2022 hemodynamic definition of PAH (mean pulmonary arterial pressure (mPAP) >20 mmHg, pulmonary artery wedge pressure (PAWP) ≤15 mmHg, and pulmonary vascular resistance (PVR) >2 WU) in the absence of other causes of pre-capillary PH (no significant ILD and no clinical suspicion of pulmonary or left sided heart disease as the predominant cause of PH), independent of diagnostic period and previous treatment
* Participants must be able to understand and follow trial procedures including completion of questionnaires regarding Patient Reported Outcome measures
* Participants must have access to the internet, and experience in using smartphones or other electronic devices with internet access.
* Capable of giving signed informed consent

Exclusion Criteria:

* Severe end organ disease

  1. Severe heart failure with EF < 30%
  2. End stage kidney disease with eGFR < 30 mL/min
  3. End stage lung disease with FVC < 50% or coexisting severe lung diseases (e.g., COPD (including emphysema), GOLD grade 3-4 with FEV1 <50%)
  4. In the opinion of the investigator, other clinically significant pulmonary abnormalities
* Active treatment for cancer or non-curable cancer
* Contraindications for functional assessment (6MWD and 1MSTS):

  1. Uncontrolled systemic hypertension (systolic >220 mmHg or diastolic >120 mmHg) or hypotension (systolic <90 mmHg), resting tachycardia (>130 beats per minute).
  2. Surgery, myocardial infarction/unstable angina, pneumothorax or stroke within the past 8 weeks.
  3. Severe musculoskeletal or neurological limitations preventing safe ambulation or any acute illness which might impair performance or safety in the opinion of the investigator.
* Unable to speak, write and read Norwegian
* Pregnancy or planned pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients diagnosed with systemic sclerosis-associated pulmonary arterial hypertension (SSc-PAH). Participants will be identified primarily through the Norwegian Systemic Connective Tissue Disease and Vasculitis Registry (NOSVAR) and routine in- and outpatient consultations. Additional recruitment will occur via the national rheumatic association, the OUH clinical studies webpage, and Helsenorge. Participants will attend two study visits at Oslo University Hospital (baseline and week 12). Given the rarity of SSc-PAH, broad recruitment is necessary to obtain feasibility data. The target enrollment is ~20 patients.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Home Monitoring: Patient Adherence and Compliance | From enrollment to the end of the study at 12 weeks
  Adherence and compliance will be assessed by tracking the frequency and completeness of data entries in the digital platform. This includes biweekly symptom reporting, completion of the 1-minute sit-to-stand test (1MSTS), and compliance with ECG monitoring.
Feasibility of Home Monitoring: Technical Feasibility | From enrollment to the end of the study at 12 weeks
  Technical feasibility will be evaluated based on the occurrence of technical failures, data loss, and missing entries in the home monitoring system. The frequency of reported technical issues and the ability of participants to successfully complete monitoring tasks will be recorded.
Feasibility of Home Monitoring: Agreement Between Home-Based 1MSTS and Hospital-Based 6MWD for Exercise Capacity Assessment | From enrollment to 12 weeks
  Agreement between home-based 1-minute sit-to-stand test (1MSTS) and hospital-based 6-minute walk distance (6MWD) in assessing exercise capacity will be evaluated using correlation analysis (e.g., Pearson or Spearman correlation) and Bland-Altman plots to assess agreement. A regression model may be applied to explore the predictive relationship between 1MSTS (number of repetitions) and 6MWD (distance in meters).
  Unit of Measure:
  * Primary Unit: Agreement (correlation coefficient)
  * Secondary Units: 1MSTS (number of repetitions), 6MWD (meters)
Feasibility of Home Monitoring: Agreement Between Home-Based and Hospital-Based Peripheral Oxygen Saturation (SpO₂) at Rest and Nadir During Exercise | From enrollment to 12 weeks
  Agreement between home-based and hospital-based peripheral oxygen saturation (SpO₂) at rest and the lowest (nadir) value during the tests.
  Unit of Measure: Percentage (%)
Feasibility of Home Monitoring: Agreement Between Home-Based and Hospital-Based Heart Rate Measurements at Rest, Peak Exercise, and Recovery | From enrollment to 12 weeks
  Agreement between home-based and hospital-based heart rate measurements at rest, at maximum during the tests, and one minute after the tests.
  Unit of Measure: Beats per minute (bpm)
Feasibility of Home Monitoring: Agreement Between Home-Based and Hospital-Based Borg Dyspnea Scale Scores During Exercise | From enrollment to 12 weeks
  Agreement between home-based and hospital-based Borg dyspnea scale scores during the tests.
  Unit of Measure: Borg dyspnea scale score
Feasibility of Home Monitoring: Agreement Between Home-Based and Hospital-Based Visual Analogue Scale (VAS) Scores for Dizziness and Palpitations | From enrollment to 12 weeks
  Agreement between home-based and hospital-based Visual Analogue Scale (VAS) scores for dizziness and palpitations from 0 - 10 cm with higher values indicating more symptoms.
  Unit of Measure: VAS score (range: 0-10 cm)
Feasibility of Home Monitoring: Agreement Between Home-Based and Hospital-Based NT-proBNP Measurements | From enrollment to 12 weeks
  Agreement between home-based and hospital-based NT-proBNP measurements. Unit of Measure: pg/mL

SECONDARY OUTCOMES:
Patient Satisfaction with Home Monitoring | 12 weeks
  Patient satisfaction with home monitoring will be assessed using the Client Satisfaction Questionnaire (CSQ-8), which evaluates overall satisfaction with the home monitoring system. The CSQ-8 consists of eight items, each rated on a 4-point scale, with a total score range of 8 to 32. Higher scores indicate greater satisfaction.
  Unit of Measure: CSQ-8 total score (range: 8-32)
Patient Usability, Feasibility and Impact of Home Monitoring | 12 weeks
  Usability, feasibility, and perceived impact of home monitoring will be assessed using a custom-designed questionnaire. This questionnaire evaluates:
  * Usability (ease of use, technical difficulties, and disease-related limitations affecting use)
  * Feasibility (time commitment, disruption to daily life, need for additional guidance)
  * Impact (perceived usefulness for disease management, confidence in self-care, and emotional responses such as anxiety) Responses will be recorded on Likert scales (1-5 or 1-4, depending on the item).
  Unit of Measure: Individual questionnaire item scores (Likert scale 1-5 or 1-4)
Patient Engagement with Healthcare Providers | From enrollment to the end of the study at 12 weeks
  The frequency and reasons for interactions between participants and healthcare providers related to home monitoring will be tracked. These interactions may include technical difficulties, concerns about home-monitoring results, and symptom-related consultations.
Impact of home monitoring on disease burden (EmPHasis-10 Score) | Baseline and 12 weeks
  The EmPHasis-10 questionnaire will be used to assess changes in disease burden and health-related quality of life (HRQoL) for patients with pulmonary arterial hypertension. The total score ranges from 0 to 50, with higher scores indicating worse HRQoL.
  Unit of Measure: EmPHasis-10 total score (range: 0-50)
Impact of home monitoring on functional status (mMRC dyspnea scale) | Baseline and 12 weeks
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used to assess changes in perceived breathlessness. The scale ranges from 0 to 4, with higher scores indicating greater dyspnea severity.
  Unit of Measure: mMRC score (range: 0-4)
Impact of home monitoring on symptoms (VAS symptom scales) | From enrollment to 12 weeks
  Patient-reported symptoms, including dyspnea, orthopnea, fatigue, dizziness, syncope, palpitations, chest pain, and edema will be assessed using Visual Analogue Scales (VAS, 0-10 cm), where higher values indicate more severe symptoms.
  Unit of Measure: VAS score (range: 0-10 cm)
Impact of home monitoring on systemic sclerosis disease burden (ScleroID Score) | Baseline and 12 weeks
  The EULAR Systemic Sclerosis Impact of Disease (ScleroID) questionnaire will be used to assess disease burden in patients with systemic sclerosis. The ScleroID evaluates ten health dimensions. Each dimension is rated on a numeric rating scale (NRS) from 0 to 10, where higher scores indicate greater disease impact. To calculate the total ScleroID score, each dimension's NRS score is multiplied by a predefined weight, reflecting its relative importance. The weighted scores are summed, resulting in a composite score ranging from 0 (no impact) to 10 (maximum impact).
  Unit of Measure: ScleroID total score (range: 0-10)
Impact of Home Monitoring on Health-Related Quality of Life (EQ-5D-5L Index Score) | Baseline and 12 weeks
  The EuroQol EQ-5D-5L descriptive system will be used to assess changes in health-related quality of life (HRQoL) across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale from no problems (Level 1) to extreme problems (Level 5). A country-specific value set will be used to calculate an index value, typically ranging from less than 0 (worse than death) to 1 (perfect health).
  Unit of Measure: EQ-5D-5L index score (range: <0 to 1)
Impact of Home Monitoring on Health-Related Quality of Life (EQ VAS Score) | Baseline and 12 weeks
  The EQ Visual Analogue Scale (EQ VAS) will be used to assess self-rated health status. Participants will rate their overall health on a vertical scale ranging from 0 (worst imaginable health) to 100 (best imaginable health).
  Unit of Measure: EQ VAS score (range: 0-100)
Impact of home monitoring on disability (HAQ Score) | Baseline and 12 weeks
  The Health Assessment Questionnaire Disability Index (HAQ-DI) will be used to assess changes in functional disability. The HAQ-DI evaluates functional ability across eight domains of daily activities: (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities). The total score ranges from 0 (no disability) to 3 (severe disability). The final HAQ-DI total score is the average of the highest scores in each domain, ranging from 0 (no disability) to 3 (severe disability). If assistive devices or assistance are required, the minimum score for that domain is adjusted to 2.
  Unit of Measure: HAQ-DI total score (range: 0-3)
Impact of home monitoring on anxiety and depression (HADS Score) | Baseline and 12 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess changes in emotional well-being. The HADS consists of two subscales (anxiety and depression), each ranging from 0 to 21, with higher scores indicating greater anxiety or depression.
  Unit of Measure: HADS total score (range: 0-42) and subscale scores (0-21)
PAH Progression | From enrollment to the end of the study at 12 weeks
  PAH progression will be defined using adapted SERAPHIN criteria, including: (i) death, (ii) lung transplantation, (iii) atrial septostomy, (iv) initiation of parenteral prostanoids, or (v) ≥15% decline in 6MWD from baseline plus worsening PAH symptoms (increased WHO-FC or signs of right heart failure unresponsive to oral diuretics) or initiation of a new PAH-specific therapy (oral/inhaled prostanoids, PDE-5is, ERAs, or sGCs). Progression events will be recorded retrospectively at the final study visit.
PAH Events | From enrollment to the end of the study at 12 weeks
  PAH events will be recorded as clinical worsening requiring healthcare utilization. Events include non-elective hospital admission or emergency department visits due to PAH, initiation of new PAH-specific therapy, and initiation of long-term oxygen therapy (LTOT). PAH events will be recorded retrospectively at the final study visit.
Changes in hospital-based clinical measures: Change in WHO Functional Class (WHO-FC) from baseline to 12 weeks | Baseline and 12 weeks
  Changes in WHO Functional Class (WHO-FC) will be assessed to evaluate changes in symptom severity and functional capacity in pulmonary hypertension. WHO-FC is categorized as:
  * Class I: No limitation of physical activity
  * Class II: Mild limitation
  * Class III: Marked limitation
  * Class IV: Unable to perform physical activity without symptoms Unit of Measure: WHO-FC classification (Ordinal scale: I-IV)
Changes in hospital-based clinical measures: Change in 6-Minute Walk Distance (6MWD) from baseline to 12 weeks | Baseline and 12 weeks
  The 6-minute walk distance (6MWD) test measures changes in exercise capacity. The total distance walked (in meters) over 6 minutes will be recorded.
  Unit of Measure: Distance in meters (m)
Changes in hospital-based clinical measures: Change in 1-Minute Sit-to-Stand Test (1MSTS) from baseline to 12 weeks | Baseline and 12 weeks
  The 1-minute sit-to-stand test (1MSTS) will assess changes in functional capacity by measuring the number of times a participant can stand up from a chair in 1 minute.
  Unit of Measure: Number of repetitions
Changes in hospital-based clinical measures: Change in Pulmonary Function Tests (PFTs) from baseline to 12 weeks | Baseline and 12 weeks
  Pulmonary function tests (PFTs) will assess changes in lung function by measuring:
  * Forced Vital Capacity (FVC, % predicted)
  * Diffusing capacity of the lung for carbon monoxide (DLCO, % predicted) Unit of Measure: Percentage of predicted value (% predicted)
Changes in hospital-based clinical measures: Change in NT-proBNP Levels from baseline to 12 weeks | Baseline and 12 weeks
  Changes in NT-proBNP levels will be assessed as a biomarker for cardiac function and disease progression.
  Unit of Measure: NT-proBNP concentration (pg/mL)
Changes in hospital-based clinical measures: Change in risk stratification score (ESC/ERS Four-Strata Model) from baseline to 12 weeks | Baseline and 12 weeks
  Changes in risk stratification will be assessed using the ESC/ERS four-strata model, which categorizes patients based on the mean score into:
  * Low risk (<1.50)
  * Intermediate-low risk (1.50-2.49)
  * Intermediate-high risk (2.50-3.49)
  * High risk (≥3.50) The classification is based on cut-off levels of WHO Functional Class (WHO-FC), 6-minute walk distance (6MWD), and NT-proBNP. Each parameter is graded 1 to 4, with the mean score defining the risk category. The model estimates 1-year mortality ranging from 0-3% (low risk) to >20% (high risk).
  Unit of Measure: Risk category (low/intermediate-low/intermediate-high/high)
Changes in Home-Based Clinical Measures | From enrollment to the end of the study at 12 weeks
  Changes in home-based clinical measures from baseline to week 12, focusing on 1-minute sit-to-stand test (1MSTS) performance over time.
Agreement Between Home-Based and Hospital-Based Risk Stratification: Determination of 1MSTS cut-offs for risk stratification based on 6MWD | From enrollment to 12 weeks
  This outcome will determine cut-off values for the 1-minute sit-to-stand test (1MSTS) that correspond to established 6-minute walk distance (6MWD) thresholds used in the ESC/ERS four-strata risk stratification model. The optimal 1MSTS cut-offs will be determined using receiver operating characteristic (ROC) curve analysis and Youden's index to identify thresholds corresponding to established 6MWD cut-off values. Correlation and regression analyses will also be used to assess the relationship between 1MSTS and 6MWD
  * Primary Unit: 1MSTS cut-off values (number of repetitions)
  * Reference Unit: 6MWD (meters)
Agreement Between Home-Based and Hospital-Based Risk Stratification: Agreement between home-based and hospital-based ESC/ERS four-strata risk stratification | From enrollment to 12 weeks
  This outcome will assess the agreement between home-based risk stratification (mMRC, 1MSTS, NT-proBNP) and hospital-based risk stratification (WHO-FC, 6MWD, NT-proBNP) using the ESC/ERS four-strata model. Patients will be categorized based on the mean score into:
  * Low risk (<1.50)
  * Intermediate-low risk (1.50-2.49)
  * Intermediate-high risk (2.50-3.49)
  * High risk (≥3.50)
  Risk classification for home-based measures will follow:
  * mMRC vs. WHO-FC: The mMRC 0-4 scale will be mapped to the WHO-FC I-IV scale based on established correlations from the COMPERA 2.0 model (mMRC 0-1 = WHO-FC I-II, mMRC 2-3 = WHO-FC III, mMRC 4 = WHO-FC IV).
  * NT-proBNP: Same cut-off values will be used for home-sampled and hospital-drawn blood.
  * 1MSTS vs. 6MWD: Cut-off values will be determined based on findings from Outcome Measure 29.
  Unit of Measure: Risk category (low/intermediate-low/intermediate-high/high)
Reproducibility of Home-Based Measures | From enrollment to the end of the study at 12 weeks
  The reproducibility of home-based measures will be assessed by comparing patient-reported mMRC vs. physician-reported WHO-FC to evaluate inter-rater agreement in functional classification and home-based 1MSTS vs. hospital-based 1MSTS to assess reproducibility across different settings.
Heart Rhythm Monitoring (ECG 247 Smart Heart Sensor) | One-week monitoring during the 12-week study period
  Home ECG monitoring will be used to assess the frequency and type of rhythm disturbances, daytime vs. nighttime heart rate (HR), heart rate variability (HRV), and correlation of HR/HRV with hospital-based measures, risk stratification, and PAH progression.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Maria Hoffmann-Vold, MD, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
The individual patient data of this study will not be publicly available as they contain information that could compromise the privacy of research participants and may be subject to ongoing research as long as the research project is ongoing. The original data will be available from the corresponding authors of subsequent publications upon reasonable request, except where restricted by GDPR liabilities.

REFERENCES:
- See also: Study information page on the Oslo University Hospital (OUH) website. — https://www.oslo-universitetssykehus.no/kliniske-studier/hjemmebasert-sykdomsoppfolging-av-pulmonal-arteriell-hypertensjon-ved-systemisk-sklerose/